CLINICAL TRIAL: NCT02250170
Title: A Phase 1, Open-label, Non-Randomized, Dose Escalation Trial to Evaluate Safety and Biomarker of OPB-111077 in Subjects With Advanced Solid Tumor
Brief Title: Safety and Biomarker of OPB-111077 in Subjects With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 317-KOA-1401i
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-111077 (Experimental): Tablet, Oral, 300mg/500mg/700mg/900mg 4 days-on & 3 days-off (21 days=1cycle)
  Interventions: Drug: OPB-111077

INTERVENTIONS:
Drug: OPB-111077 — Tablet, Oral, 300mg/500mg/700mg/900mg 4 days-on & 3 days-off (21 days=1cycle)

SUMMARY:
This open-label, non-randomized trial will comprise of 2 parts. A dose escalation part will characterize the safety, biomarker and pharmacokinetics of OPB-111077 in advanced solid tumor. Subsequently, an expansion part will further evaluate the biomarker, safety, pharmacokinetics and antitumor activity of OPB-111077 in selected tumor types.

DETAILED DESCRIPTION:
This trial is designed to determine the safety, tolerability, maximum tolerated dose and recommended dose of OPB-111077 administered orally 4-days on and 3-days off (3 weeks/cycle) to subjects with advanced solid tumor in the dose escalation part so that biomarkers, efficacy, and others can be evaluated at the recommended dose in an expeditious manner in the expansion part. The dose escalation part employs a 3+3 escalation design as a standard dose escalation design for a small sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically and/or cytologically confirmed advanced solid tumor
2. Patients who were refractory to standard therapy or for which there are no standard treatment options available
3. Age 20 to 80 years at the time of informed consent
4. Patients who, together with their partner, are willing and capable of using an appropriate method of contraception throughout the trial period and until at least 12 weeks after final IMP administration
5. Patients informed of the diagnosis of advanced solid tumor who are fully informed about the content of the study by the investigator or subinvestigator using the specified written consent form and other written explanation, and give written consent to participate in the study of their free will
6. Patients who are able to take oral medication

Exclusion Criteria:

1. Patients with symptomatic brain metastases
2. Patients who have not recovered from any prior therapy related toxicity deemed to be clinically significant at study entry, except for the test item defined in inclusion criteria.
3. Patients with active infections needing whole body therapy
4. Patients with positive hepatitis B surface (HBs) antigen or positive hepatitis C virus (HCV) antibody
5. Patients with positive human immunodeficiency virus (HIV) antibody
6. Patients with uncontrollable cardiac diseases
7. Patients with uncontrollable pain by analgesic drugs
8. Patients with a history of organ transplantation
9. Patients who have received another IMP
10. Patients who are pregnant, possibly pregnant, or lactating
11. Patients otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 21 days
  Number of participants with Adverse Events
Maximum tolerated dose | 21 days
  The highest dose that does not lead to discontinuation of dose escalation
Biomarker of OPB-111077 | 21 days
  Change from baseline on predictable biomarker specified in the protocol

SECONDARY OUTCOMES:
Tumor response measured by RECIST(Response Evaluation Criteria in Solid Tumor) 1.1 Assessment | 3~18 weeks depending on tumor response
  Tumor response measured by RECIST(Response Evaluation Criteria in Solid Tumor) 1.1 Assessment will be conducted at Screening, end of Cycle 1, end of Cycle 2, end of every 2 cycles thereafter, at the final study visit.
Pharmacokinetics (PK) properties of OPB-111077 and its metabolites. | 21 days
  The following PK parameters (Cmax (maximum observed concentration), AUC(area uder the concentration time curve from zero), tmax (Time to maximum plasma concentration), etc.) will be determined using a non-compartmental methods.

CONTACTS AND LOCATIONS:
Overall Officials: Doyoun Oh, MD, Principal Investigator — Seoul National University Hospital; Jeehyun Kim, MD, Principal Investigator — Seoul National University Bundang Hospital; Sungbae Kim, MD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul